CLINICAL TRIAL: NCT05894733
Title: The Effects of Frequent Follow up on Compliance in Patients Receiving PAP Therapy Due to OSA
Brief Title: The Effects of Frequent Follow up on Compliance in Patients Receiving PAP Therapy Due to OSA (Pap: Positive Airway Pressure, OSA: Obstructive Sleep Apnea )
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Makbule Özlem Akbay, medical doctor, Istanbul Sureyyapasa Chest Diseases and Chest Surgery Training and Research Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 1
Record Dates: First submitted 2023-05-26; First posted 2023-06-08 (Actual); Last update posted 2023-06-08 (Actual); Status verified 2023-06

CONDITIONS: Patient Compliance; Sleep Disorder; Obstructive Sleep Apnea of Adult
MeSH Terms: conditions — Patient Compliance; Sleep Wake Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 (Other): 1: The first group was called by phone on the 15th day to ask if there were any complaints or problems with the device. Sequentially, they were called for controls at the end of the first, third, and sixth months.
  Interventions: Other: study group
- 2 (Other): 2:The second group was accepted as the control group, following our clinic's standard procedure in the first and sixth months
  Interventions: Other: control group

INTERVENTIONS:
Other: study group — Calling with phone frequently(15.th day, 1 month , 3 month, 6 month ) and face to face interwiew on first, 3 th and 6th month
  Arms: 1
Other: control group — first and sixth month face to face interwiew
  Arms: 2

SUMMARY:
The investigators planned to investigate the effect of close monitoring on compliance and the factors affecting compliance among patients receiving PAP treatment due to OSA.This study was a single-center, prospective, randomized, controlled study approved by the hospital's ethics committee.One hundred twenty-eight patients were randomized as group one or two as group 1 is the study and group 2 is the control group. The first group was called by phone on the 15th day to ask if there were any complaints or problems with the device. Sequentially, they were called for controls at the end of the first, third, and sixth months.

The second group was accepted as the control group, following our clinic's standard procedure in the first and sixth months. The patients who came to the control were asked if there were any problems with the device and any difficulties in use, and they were again informed about the devices and masks.

ELIGIBILITY:
Inclusion Criteria:, .newly diagnosed OSA with PSG , and underwent PAP titration

Exclusion Criteria:

. unfollowed patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
follow-up | 1 year
  Short-term compliance( mean duration time to use CPAP therapy) was measured during the first follow-up, and long-term compliance was measured during the last follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: makbule özlem akbay, md, Principal Investigator — sureyyapasa chest diseases center
Locations (1):
- Makbule Özlem, Maltepe, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No